CLINICAL TRIAL: NCT02000219
Title: A Phase 2 Open-label Multi-centre Study to Evaluate the Efficacy and Safety of Oxabact® to Reduce Plasma Oxalate in Subjects With Primary Hyperoxaluria Who Are on Dialysis
Brief Title: Study to Evaluate the Efficacy and Safety of Oxabact (OC5) in Primary Hyperoxaluria Patients Who Are on Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OxThera (Industry)
Collaborators: FP7-SME-2013 Research for the benefit of SMEs program (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC5-OL-01
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-10

CONDITIONS: Primary Hyperoxaluria
Keywords: hyperoxaluria; oxalate; PH; dialysis
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxabact OC5 capsule (Experimental): This is an open-label study so all patients will receive the active drug product, Oxalobacter formigenes, OC5. This will be administered as an enteric-coated capsules twice daily for 6 weeks of treatment.
  In Germany, the protocol has been amended such that patients can receive OC5 for a further 3 year of continued treatment after the initial part of the study.
  Interventions: Biological: Oxalobacter formigenes

INTERVENTIONS:
Biological: Oxalobacter formigenes — The dose will be (not less than) NLT ≥1E+09 colony forming units (CFU) twice daily. The dose (an enteric-coated capsule) will be administered orally with breakfast and dinner.
  Other Names: Oxabact; OC5

SUMMARY:
The purpose of this study is to determine if Oxalobacter formigenes is effective at lowering plasma oxalate levels in patients with primary hyperoxaluria who are on dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (as applicable for the age of the subject). An appendix to the informed consent will be signed by patients continuing on treatment after week 14.
2. Male or female subjects ≥ 2 years of age. Subjects have to be able to swallow size 4 capsules twice daily for 6 weeks, or use a gastric tube that allows for administration of size 4 capsules.
3. A diagnosis of PH (as determined by standard diagnostic methods).
4. Patient should be on a stable dialysis regimen for at least two weeks before baseline.
5. Pre-dialysis plasma oxalate ≥40 micromole/L.
6. Patients receiving vitamin B6 must be receiving a stable dose for at least 3 months prior to screening and must remain on the stable dose during the study. Patients not receiving vitamin B6 at study entry must be willing to refrain from initiating vitamin B6 during study participation.

   Exclusion Criteria:
7. Inability to swallow size 4 capsules twice daily for 6 weeks or using a gastric tube not suited for administration of size 4 capsules via the tube.
8. Ongoing treatment with immunosuppressive medication.
9. The existence of secondary hyperoxaluria, e.g. hyperoxaluria due to bariatric surgery or chronic gastrointestinal diseases such as cystic fibrosis, chronic inflammatory bowel disease and short-bowel syndrome.
10. Use of antibiotics to which O. formigenes is sensitive, including current antibiotic use, or antibiotics use within 14 days of initiating study medication.
11. Current treatment with a separate ascorbic acid preparation. Standard of care vitamin supplement for patients on dialysis is allowed.
12. Pregnancy.
13. Women of childbearing potential who are not using adequate contraceptive precautions. Sexually active females, unless surgically sterile or at least 2 years post-menopausal, must be using a highly effective contraception (including oral, transdermal, injectable, or implanted contraceptives, IUD, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 30 days prior to the first dose of OC5 and must agree to continue using such precautions during the clinical study.
14. Presence of a medical condition that the Investigator considers likely to make the subject susceptible to adverse effect of study treatment or unable to follow study procedures.
15. Participation in any study of an investigational product, biologic, device, or other agent within 30 days prior to the first dose of OC5 or not willing to forego other forms of investigational treatment during this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gesa Schalk, M.D., Principal Investigator — University of Bonn
Locations (1):
- Universitätsklinikum Bonn, Department of Paediatric Nephrology, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxabact OC5 Capsule: This is an open-label study so all patients will receive the active drug product, Oxalobacter formigenes, OC5. This will be administered as an enteric-coated capsules twice daily for 6 weeks of treatment.
  In Germany, the protocol has been amended such that patients can receive OC5 for a further 3 year of continued treatment after the initial part of the study.
  Oxalobacter formigenes: The dose will be (not less than) NLT ≥1E+09 colony forming units (CFU) twice daily. The dose (an enteric-coated capsule) will be administered orally with breakfast and dinner.
Period: 14-Week Study Period
Arm/Group | Oxabact OC5 Capsule
Started | 12
Completed | 9
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Underwent transplantation | 1
Period: Continuation Period
Arm/Group | Oxabact OC5 Capsule
Started (One patient chose not to enter the continuation period, and returned to their home country) | 8
Completed | 3
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Had liver transplant | 2
Not completed — Non-compliance with study drug | 2

BASELINE CHARACTERISTICS:
Population: Patients with primary hyperoxaluria (PH) who are on dialysis
Arm/Group | Oxabact OC5 Capsule
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  France | 1
  Germany | 11
Primary hyperoxaluria Type I [Count of Participants; unit: Participants] — Primary Hyperoxaluria is the result of rare genetic mutations. The three main types of primary hyperoxaluria are the result of different gene deficiencies.
  Primary Hyperoxaluria Type I is the result of mutations in the AGXT gene (alanine-glyoxylate aminotransferase).
  Primary Hyperoxaluria Type II is the result of mutations in the GRHPR gene (glyoxylate reductase-hydroxypyruvate reductase)
  Participants | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Pre Dialysis Plasma Oxalate (Total Plasma Oxalate) Level During Treatment With OC5 Compared With Baseline.
Description: Total plasma oxalate measured in umol/L
Time Frame: Baseline (average of week 2 & 4 pretreatment); treatment weeks 6, 8 & 10 (on treatment 2, 4, & 6 weeks); off treatment weeks 12 & 14 (2 & 4 weeks off treatment); patients were then eligible for treatment up to 3 years & oxalate was measured every 6 months
Population: Data presented by visit for patients completing each visit
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Oxabact OC5 Capsule
Number analyzed (Participants) | 12
μmol/L
  Baseline value (average of week 2 and 4 pretreatment) | 147.57 (39.63)
  2 week treatment change from baseline | 11.34 (2.68)
  4 week treatment change from baseline: number analyzed (Participants) | 11
  4 week treatment change from baseline | 7.46 (26.93)
  6 week treatment change from baseline: number analyzed (Participants) | 10
  6 week treatment change from baseline | -5.68 (21.02)
  2 week off treatment change from baseline: number analyzed (Participants) | 9
  2 week off treatment change from baseline | -4.56 (18.23)
  4 week off treatment change from baseline: number analyzed (Participants) | 9
  4 week off treatment change from baseline | -8.41 (19.26)
  continued treatment 24 weeks change from baseline: number analyzed (Participants) | 8
  continued treatment 24 weeks change from baseline | -35.99 (42.60)
  continued treatment 52 weeks change from baseline: number analyzed (Participants) | 6
  continued treatment 52 weeks change from baseline | -33.99 (34.78)
  continued treatment 76 weeks change from baseline: number analyzed (Participants) | 6
  continued treatment 76 weeks change from baseline | -28.04 (38.45)
  continued treatment 104 weeks change from baseline: number analyzed (Participants) | 5
  continued treatment 104 weeks change from baseline | -67.36 (47.77)
  continued treatment 128 weeks change from baseline: number analyzed (Participants) | 4
  continued treatment 128 weeks change from baseline | -46.25 (26.90)
  continued treatment 156 weeks change from baseline: number analyzed (Participants) | 3
  continued treatment 156 weeks change from baseline | -44.65 (54.75)

2. Secondary Outcome: Change in Pre Dialysis Plasma Oxalate (Free Plasma Oxalate) Level During Study Compared With Baseline.
Description: Comparison of free plasma oxalate compared to the four week baseline period.
Time Frame: as for outcome 1
Population: Patients completing each study visit are included
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Oxabact OC5 Capsule
Number analyzed (Participants) | 12
μmol/L
  Baseline: number analyzed (Participants) | 8
  Baseline | 106.91 (35.50)
  Change from baseline at the end of six weeks of treatment: number analyzed (Participants) | 8
  Change from baseline at the end of six weeks of treatment | 1.59 (18.77)
  Change from baseline 4 weeks after treatment for 6 weeks: number analyzed (Participants) | 7
  Change from baseline 4 weeks after treatment for 6 weeks | -6.50 (17.31)
  Change from baseline at 24 weeks: number analyzed (Participants) | 8
  Change from baseline at 24 weeks | -10.17 (15.27)
  Change from baseline at 52 weeks: number analyzed (Participants) | 5
  Change from baseline at 52 weeks | 2.52 (13.79)
  Change from baseline at 76 weeks: number analyzed (Participants) | 5
  Change from baseline at 76 weeks | -17.47 (13.71)
  Change from baseline at 104 weeks: number analyzed (Participants) | 4
  Change from baseline at 104 weeks | -47.29 (30.46)
  Change from baseline at 128 weeks: number analyzed (Participants) | 3
  Change from baseline at 128 weeks | -38.54 (10.59)
  Change from baseline at 156 weeks: number analyzed (Participants) | 2
  Change from baseline at 156 weeks | -5.36 (20.99)

3. Secondary Outcome: Change in Left Ventricular Ejection Fraction From Baseline.
Description: Mean left ventricular ejection fraction measured as a percentage. Reference range 55-70%.
Time Frame: At baseline and approximately every 6 months throughout the 3 year continued treatment.
Population: Data presented for patients with baseline and visit values recorded
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Oxabact OC5 Capsule
Number analyzed (Participants) | 12
Percent
  Baseline: number analyzed (Participants) | 10
  Baseline | 50.20 (10.26)
  Week 24: number analyzed (Participants) | 7
  Week 24 | 59.43 (4.08)
  Week 52: number analyzed (Participants) | 6
  Week 52 | 59.83 (5.85)
  Week 80: number analyzed (Participants) | 5
  Week 80 | 59.60 (5.18)
  Week 104: number analyzed (Participants) | 5
  Week 104 | 59.40 (5.94)
  Week 128: number analyzed (Participants) | 4
  Week 128 | 58.00 (2.16)
  Week 156: number analyzed (Participants) | 3
  Week 156 | 58.67 (7.57)

4. Secondary Outcome: Speckle Tracking Echocardiography
Description: Global longitudinal strain (GLS), which measures the maximal shortening of myocardial longitudinal length during systole compared to the resting length in diastole. The normal range for GLS is considered to be < -18%.
Time Frame: At baseline and approximately every 6 months throughout the 3 year continued treatment.
Population: Data presented for patients completing analyses
Measure: Mean (Standard Deviation); unit: percentage of myocardial length change
Arm/Group | Oxabact OC5 Capsule
Number analyzed (Participants) | 9
percentage of myocardial length change
  Baseline value | -17.37 (5.30)
  Week 24: number analyzed (Participants) | 6
  Week 24 | -19.15 (2.52)
  Week 52: number analyzed (Participants) | 6
  Week 52 | -18.29 (3.27)
  Week 80: number analyzed (Participants) | 5
  Week 80 | -19.53 (1.65)
  Week 104: number analyzed (Participants) | 5
  Week 104 | -19.99 (2.96)
  Week 128: number analyzed (Participants) | 4
  Week 128 | -19.60 (1.73)
  Week 156: number analyzed (Participants) | 3
  Week 156 | -18.52 (1.65)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through last follow up visit, up to 3 years
Arm/Group | Oxabact OC5 Capsule
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 7/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxabact OC5 Capsule (N=12)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (2)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (2)
Device related infection (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxabact OC5 Capsule (N=12)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (12)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (7)
Dialysis device insertion (Surgical and medical procedures) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator may not publish the results of their cohort of subjects until the full study has been submitted for publication. They may not submit for publication or present the results of this study without allowing OxThera 30 days in which to review and comment on the pre-publication manuscript. The investigator may not submit the results of the study for publication without the prior consent of OxThera, unless the review period has passed and there has been no reaction from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02000219/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02000219/SAP_001.pdf